CLINICAL TRIAL: NCT03385785
Title: Ventriculo-arterial Coupling Modification Evaluated by PRAM (Pressure Recording Analytical Method) in the Aortic Stenosis Treated by TAVI (Transcatheter Aortic Valve Implantation)
Brief Title: Ventriculo-arterial Coupling Modification Evaluated by PRAM During TAVI Procedure
Acronym: PRAM-TAVI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2017/PRAMTAVI-FRITZ/YB
Record Dates: First submitted 2017-10-24; First posted 2017-12-29 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-09

CONDITIONS: Aortic Valve Stenosis; Ventricular Dysfunction, Left
Keywords: Transcatheter aortic valve replacement; Pressure Recording Analytical Method; Ventriculo-arterial coupling; Monitoring; Hemodynamic
MeSH Terms: conditions — Aortic Valve Stenosis; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Calcified aortic stenosis is the most frequent valvulopathy in Europe and North America. Aortic stenosis is an obstacle to the ejection of blood from the left ventricle to the aorta and leads to morphological changes in the left ventricle and hemodynamic modifications.

Intrinsic ventricular performance can be characterized using three parameters:

* Ventricular elastance (Ees for End Systolic Elastance) which represents the index of ventricular contractility independently of the load.
* Arterial elastance (Ea for Arterial Elastance) which represents the post-load
* The ventriculo-arterial coupling index (Ees / Ea) which represents energy efficiency.

For patients with high surgical risk (EuroSCORE II> 6), TAVI (Transcatheter Aortic Valve Implantation) is recommended for aortic valve replacement. Many complications may occur after TAVI (haemorrhagic, embolic, renal, myocardial ischemia). Post-TAVI complications may also be cardiac decompensation of the underlying cardiac disease to cardiogenic shock. However, literature on left ventricular performance after aortic valvular replacement is poor because of the difficulty and invasiveness of the analysis involved.

Cardiac energy analysis plays an additional role in understanding the clinical patients conditions. On this point, cardiac energy modifications, based on ventriculo-arterial coupling, could be indicators of cardiac function. Two methods (ultrasound and pulse contour) are used to understand and explore the ventriculo-arterial coupling, preload, postload, contractility and hemodynamic changes interactions.

Echocardiography allows the Ees / Ea and SW / PVA (Stoke work/ pressure-volume area) ratios mesurements. PRAM (Pressure Recording Analytical Method) through the MostCare® monitor, gives common hemodynamic parameters and more specific parameters such as arterial elastance (Ea) cardiac cycle efficiency (CCE), dP / dt. Cardiac cycle efficiency (CCE) is an exclusive variable that describes the hemodynamic performance in terms of energy expenditure in the patient being followed.

TAVI procedure is an acute model of ventriculo-arterial coupling modification by treatment of the ventricular ejection obstacle. The PRAM method evaluates the ventriculo-arterial coupling. The aim of our study is to evaluate by PRAM the changes in cardiac energy variables before and after aortic valve replacement by TAVI

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* elective TAVI intervention with femoral access
* consent

Exclusion Criteria:

* permanent arrhythmias
* pacemaker dependency
* moderate to severe mitral or tricuspid valve regurgitation
* intracardiac shunt

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patients hospitalized for TAVI
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Transcatheter aortic valve implantation (TAVI) impact on cardiac energy performance | Change from baseline CCE at 30 minutes after transcatheter aortic valve implantation
  Mesurement of the cardiac cycle efficency (CCE) by PRAM method (Pressure Recording Analytical Method)

SECONDARY OUTCOMES:
Echocardiographic cardiac energy performance modification after transcatheter aortic valve implantation | Change from baseline at 24 hours after transcatheter aortic valve implantation
  Echocardiography explorations (end diastolic diameter, end systolic diameter, diastolic wall thickness, systolic wall thickness, end diastolic volume, end systolic volume, percent fractional shortening, percent ejection fraction)
Myocardial ischemia risk | Change from baseline at 24 hours after transcatheter aortic valve implantation
  Buffington index (calculated as : mean arterial pressure / heart rate)
Myocardial ischemia | Change from baseline at 24 hours after transcatheter aortic valve implantation
  Serum troponin level

CONTACTS AND LOCATIONS:
Overall Officials: Caroline FRITZ, MD, Principal Investigator — Central Hospital, Nancy, France
Locations (1):
- FRITZ, Nancy, France